CLINICAL TRIAL: NCT02857283
Title: Human Biological Responses to Low Level Ozone
Acronym: SNOZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Environmental Protection Agency (EPA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 15-2677
Record Dates: First submitted 2016-06-27; First posted 2016-08-05 (Estimated); Results first posted 2020-04-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Environmental Exposure; Nasal Inflammation
Keywords: Air pollution; Air pollutant exposure; Ozone
MeSH Terms: interventions — Ozone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Filtered Air, then Ozone (Experimental): Participants in this arm will first receive filtered clean air followed by ozone
  Interventions: Other: Ozone; Other: Filtered Air; Device: Health and Exposure Tracker (HET)
- Ozone, then Filtered Air (Experimental): Participants in this arm will first receive ozone followed by filtered clean air
  Interventions: Other: Ozone; Other: Filtered Air; Device: Health and Exposure Tracker (HET)

INTERVENTIONS:
Other: Ozone — Participants will be exposed to a concentration of ozone for 6.5 hours at a concentration that varies 0.06 to 0.08
Other: Filtered Air — Participants will be exposed to filtered clean air
Device: Health and Exposure Tracker (HET) — Ozone and heart rate tracker

SUMMARY:
To investigate if low level ozone exposure will cause measurable inflammation in nasal cells.

DETAILED DESCRIPTION:
Air pollutants including ozone have been implicated in affecting health outcomes. In particular, high level ozone exposure has been shown to affect pulmonary function and cause pulmonary inflammation. Troubling community-based work has implicated high ozone levels as being correlated with increased pediatric asthma emergency room visits. Because of adverse health effects, EPA standards for safe ozone levels have been set, currently at 0.07 ppm. Still, it is estimated that 100 million Americans live in areas where ozone levels periodically remain above the EPA standard. And while this EPA standard had been set based on available data, it remained unclear at the time whether naturalistic low-level ozone exposure, such as fluctuations between 0.06-0.08 ppm throughout the day, might affect health as well.

This group previously examined lung function and inflammatory response in adults exposed to low-level ozone, 0.06 ppm exposure for 6.6 hours, while undergoing intermittent moderate exercise. The investigators found that in response to low-level ozone exposure (0.06 ppm) with exercise, lung function declines and neutrophilic airway inflammation is observed. What remains unclear, is whether low-level ozone alone - without exercise - will cause similar health effects.

To mimic exposure to ozone on a typical summer day in a polluted city, the investigators will expose subjects to a varying level of ozone, form 0.06 ppm to 0.08 ppm, rather than a constant 0.07ppm. The variation from 0.06ppm to 0.08ppm, then back to 0.06ppm will occur each hour.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18 and 50 years of age.
* Vital signs within normal limits on admission to the study: Peripheral oxygen saturation (SpO2) > 94%, systolic blood pressure between 150-90 mm Hg, diastolic blood pressure between 100-60 mm Hg, afebrile.
* Forced Expiratory Volume (FEV1) of at least 80% of predicted.

Exclusion Criteria:

* Any chronic medical condition considered by the PI as a contraindication to the exposure study, including significant cardiovascular disease, diabetes requiring medication, chronic renal disease, chronic thyroid disease, or kidney disease.
* Use of systemic or inhaled steroids.
* Use of NSAID or aspirin within 7days of each study visit, and inability to withhold these medications prior to each session of the study.
* Pregnant or nursing women
* Use of cigarettes or other inhaled nicotine products within the past year, or more than a lifetime 5 pack year history of cigarette smoking.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-04-22 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David B Peden, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Center for Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Peden DB, Setzer RW Jr, Devlin RB. Ozone exposure has both a priming effect on allergen-induced responses and an intrinsic inflammatory action in the nasal airways of perennially allergic asthmatics. Am J Respir Crit Care Med. 1995 May;151(5):1336-45. doi: 10.1164/ajrccm.151.5.7735583.
- [Background] Little, R. J. and Rubin, D. B. (2014). Statistical analysis with missing data. John Wiley & Sons.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 17 participants were screened between April 22, 2017 and May 1, 2019. Participants were recruited from a database of subjects at the Center for Environmental Medicine, Asthma and Lung Biology.
Pre-assignment Details: Two participants did not meet inclusion criteria, and 1 withdrew before undergoing the second exposure. All participants were free from acute illness
Groups:
- Filtered Air; Then Ozone: Participants were exposed to filtered clean air for 6.5 hours, and after a minimum of a 2-week washout, they returned and were exposed to 0.06-0.08 Parts Per Million (PPM) ozone for 6.5 hours. All participants wore a Health and Exposure Tracker (HET): Ozone and heart rate tracker during both exposures.
- Ozone; Then Filtered Air: Participants were exposed to 0.06-0.08 PPM ozone for 6.5 hours, and after a minimum of a 2-week washout, they returned and were exposed to filtered clean air for 6.5 hours. All participants wore a Health and Exposure Tracker (HET): Ozone and heart rate tracker during both exposures.
Period: First Exposure
Arm/Group | Filtered Air; Then Ozone | Ozone; Then Filtered Air
Started | 8 | 7
Completed | 7 | 7
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Washout (2 Weeks)
Arm/Group | Filtered Air; Then Ozone | Ozone; Then Filtered Air
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Second Exposure
Arm/Group | Filtered Air; Then Ozone | Ozone; Then Filtered Air
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who completed the study; one participant who dropped out after the first exposure (Filtered Air) is excluded
Groups:
- Filtered Air; Then Ozone: Participants were exposed to filtered clean air for 6.5 hours, and after a minimum of a 2-week washout, they returned and were exposed to 0.06-0.08 PPM ozone for 6.5 hours. All participants wore a Health and Exposure Tracker (HET): Ozone and heart rate tracker during both exposures
- Total: Total of all reporting groups
Arm/Group | Filtered Air; Then Ozone | Ozone; Then Filtered Air | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Full Range); unit: years] | 28.8 [22.4 to 38.0] | 35.47 [31.0 to 40] | 31.22 [22.4 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 5 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — United States, Residents of North Carolina, all within 50 miles of Chapel Hill
  Participants
    United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in % Polymorphonuclear Leukocytes (PMN) in Nasal Lavage Fluid Immediately Post-Exposure From Baseline
Description: Participants will be exposed to either filtered air (FA), then ozone (O3), or O3, then FA. Nasal lavage fluid (NLF) will be collected from participants at a baseline visit within two weeks prior to each exposure, and at the following time points for each exposure: immediately after exiting the exposure chamber, and at 24 hours after the exposure.
  The % PMN as a percentage of total inflammatory cells (total of monocytes and macrophages, PMN, eosinophils, basophils, lymphocytes, and bronchial epithelial cells) will be determined in each NLF collection by differential counts of cells on cytospin slides. The change in the values from baseline to immediately Post-Exposure will be calculated for each participant for each exposure. Values will be compared between FA and O3.
Time Frame: Baseline, immediately post-exposure
Population: Only 5 participants had paired pre and immediately post-filtered air exposure samples and only 3 had paired pre and immediately post-ozone exposure samples of adequate quality for analysis. Only 1 participant had paired samples from both exposure periods. The remainder of samples were of poor quality and contained insufficient cells for analysis.
Measure: Mean (Standard Error); unit: percent PMNs in nasal lavage fluid
Groups:
- Filtered Air: Participants will be exposed to filtered clean air for 6.5 hours
- Ozone: Participants will be exposed to a concentration of ozone for 6.5 hours at a concentration that varies 0.06 to 0.08 Parts Per Million (PPM)
Arm/Group | Filtered Air | Ozone
Number analyzed (Participants) | 5 | 3
percent PMNs in nasal lavage fluid | -1.02 (10.57) | -6.8 (6.75)

2. Primary Outcome: Change in % Polymorphonuclear Leukocytes (PMN) in Nasal Lavage Fluid 24 Hours Post-Exposure From Baseline
Description: Participants will be exposed to either filtered air (FA), then ozone (O3), or O3, then FA. Nasal lavage fluid (NLF) will be collected from participants at a baseline visit within two weeks prior to each exposure, and at the following time points for each exposure: immediately after exiting the exposure chamber, and at 24 hours after the exposure.
  The % PMN as a percentage of total inflammatory cells (total of monocytes and macrophages, PMN, eosinophils, basophils, lymphocytes, and bronchial epithelial cells) will be determined in each NLF collection by differential counts of cells on cytospin slides. The change in the values from baseline to 24 hours Post-Exposure will be calculated for each participant for each exposure. Values will be compared between FA and O3.
Time Frame: Baseline, 24 hours post-exposure
Population: Only 5 participants had paired pre and 24h post-filtered air exposure samples and only 3 had paired pre and 24h post-ozone exposure samples of adequate quality for analysis. Only 1 participant had paired samples from both exposure periods. The remainder of samples were of poor quality and contained insufficient cells for analysis.
Measure: Mean (Standard Error); unit: percent PMNs in nasal lavage fluid
Groups:
- Ozone: Participants will be exposed to a concentration of ozone for 6.5 hours at a concentration that varies 0.06 to 0.08 PPM
Arm/Group | Filtered Air | Ozone
Number analyzed (Participants) | 5 | 3
percent PMNs in nasal lavage fluid | 17.18 (16.76) | -27.97 (31.67)

3. Secondary Outcome: Interleukin-6 (IL-6) Concentrations in Nasal Epithelial Lining Fluid (ELF): Change Immediately Post-Exposure From Baseline
Description: Participants will be exposed to either filtered air (FA), then ozone (O3), or O3, then FA. Nasal epithelial lining (ELF) will be collected from participants at a baseline visit within two weeks prior to each exposure, and at the following time points for each exposure: immediately after exiting the exposure chamber, and at 24 hours after the exposure.
  The IL-6 concentration will be determined in each ELF sample by immunoassay. The change in IL-6 concentrations from baseline to immediately Post-Exposure will be calculated for each participant for each exposure. Values will be compared between FA and O3 to determine the effect of ozone on the production of nasal IL-6.
Time Frame: Baseline, immediately post-exposure
Population: All participants that completed the study
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Filtered Air | Ozone
Number analyzed (Participants) | 14 | 14
pg/mL | 2.28 (2.01) | 5.33 (3.19)
Statistical Analysis 1: Comparison: Filtered Air vs Ozone; Test type: Superiority; p = 0.46, ANOVA; paired

4. Secondary Outcome: % Polymorphonuclear Leukocytes (PMN) in Induced Sputum: Change 24 Hours Post-Exposure From Screening Visit
Description: Participants will be exposed to either filtered air (FA), then ozone (O3), or O3, then FA. Induced sputum will be collected from participants after inhaled hypertonic saline. Induced sputum will be collected at the screening visit within six weeks prior to the first exposure, and at 24 hours after each exposure.
  The % PMN as a percentage of total inflammatory cells (total of monocytes and macrophages, PMN, eosinophils, basophils, lymphocytes, and bronchial epithelial cells) will be determined in each induced sputum collection by differential counts of cells on cytospin slides. The change in the values from baseline to 24 hours Post-Exposure will be calculated for each participant for each exposure. Values will be compared between FA and O3.
Time Frame: Screening visit and 24 hours post-exposure
Population: Participants who produced induced sputum containing at least 60000 inflammatory cells at both the screening visit and at 24 hours after at least one exposure
Measure: Mean (Standard Error); unit: percent PMN
Arm/Group | Filtered Air | Ozone
Number analyzed (Participants) | 9 | 10
percent PMN | 12.04 (5.22) | 21.86 (7.74)
Statistical Analysis 1: Comparison: Filtered Air vs Ozone; Test type: Superiority; p = 0.0481, ANOVA; Paired

5. Secondary Outcome: The Percentage of Predicted Forced Expiratory Volume in One Second (% Predicted FEV1): Change Immediately Post-Exposure From Baseline
Description: Participants will be exposed to either filtered air (FA), then ozone (O3), or O3, then FA. Standard spirometry to obtain FEV1 and forced vital capacity (FVC) measurements will be done at baseline within two weeks prior to first exposure, and immediately after exiting the exposure chamber for each exposure.
  The % Predicted FEV1 will be calculated from measured versus expected values. The change in % Predicted FEV1 from baseline to immediately Post-Exposure will be calculated for each participant for each exposure. Values will be compared between FA and O3 to determine the effect of ozone on the % Predicted FEV1.
Time Frame: Baseline, immediately post-exposure
Population: All participants that completed the study
Measure: Mean (Standard Error); unit: percent predicted FEV1
Arm/Group | Filtered Air | Ozone
Number analyzed (Participants) | 14 | 14
percent predicted FEV1 | 0.79 (0.70) | -2.00 (0.70)
Statistical Analysis 1: Comparison: Filtered Air vs Ozone; Test type: Superiority; p = 0.0179, ANOVA

6. Secondary Outcome: Interleukin-6 (IL-6) Concentrations in Nasal Epithelial Lining Fluid (ELF): Change 24 Hours Post-Exposure From Baseline
Description: Participants will be exposed to either filtered air (FA), then ozone (O3), or O3, then FA. Nasal epithelial lining (ELF) will be collected from participants at baseline within two weeks prior to first exposure, and at the following time points for each exposure: immediately after exiting the exposure chamber, and at 24 hours after the exposure.
  The IL-6 concentration will be determined in each ELF sample by immunoassay. The change in IL-6 concentrations from baseline to 24 hours Post-Exposure will be calculated for each participant for each exposure. Values will be compared between FA and O3 to determine the effect of ozone on the production of nasal IL-6.
Time Frame: Baseline, 24 hours post-exposure
Population: All participants that completed the study
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Filtered Air | Ozone
Number analyzed (Participants) | 14 | 14
pg/ml | 4.15 (2.57) | 11.25 (3.56)
Statistical Analysis 1: Comparison: Filtered Air vs Ozone; Test type: Superiority; p = 0.10, ANOVA; paired

7. Secondary Outcome: Interleukin-8 (IL-8) Concentrations in Nasal Epithelial Lining Fluid (ELF): Change Immediately Post-Exposure From Baseline
Description: Participants will be exposed to either filtered air (FA), then ozone (O3), or O3, then FA. Nasal epithelial lining (ELF) will be collected from participants at baseline within two weeks prior to first exposure, and at the following time points for each exposure: immediately after exiting the exposure chamber, and at 24 hours after the exposure.
  The IL-8 concentration will be determined in each ELF sample by immunoassay. The change in IL-8 concentrations from baseline to immediately Post-Exposure will be calculated for each participant for each exposure. Values will be compared between FA and O3 to determine the effect of ozone on the production of nasal IL-8.
Time Frame: Baseline, immediately post-exposure
Population: All participants that completed the study
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Filtered Air | Ozone
Number analyzed (Participants) | 14 | 14
pg/mL | 2036.75 (1518.94) | 2939.08 (1885.08)
Statistical Analysis 1: Comparison: Filtered Air vs Ozone; Test type: Superiority; p = 0.69, ANOVA; paired

8. Secondary Outcome: Interleukin-8 (IL-8) Concentrations in Nasal Epithelial Lining Fluid (ELF): Change 24 Hours Post-Exposure From Baseline
Description: Participants will be exposed to either filtered air (FA), then ozone (O3), or O3, then FA. Nasal epithelial lining (ELF) will be collected from participants at baseline within two weeks prior to first exposure, and at the following time points for each exposure: immediately after exiting the exposure chamber, and at 24 hours after the exposure.
  The IL-8 concentration will be determined in each ELF sample by immunoassay. The change in IL-8 concentrations from baseline to 24 hours Post-Exposure will be calculated for each participant for each exposure. Values will be compared between FA and O3 to determine the effect of ozone on the production of nasal IL-8.
Time Frame: Baseline, 24 hours post-exposure
Population: All participants that completed the study
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Filtered Air | Ozone
Number analyzed (Participants) | 14 | 14
pg/mL | 3524.77 (2165.80) | 6696.56 (3032.59)
Statistical Analysis 1: Comparison: Filtered Air vs Ozone; Test type: Superiority; p = 0.27, ANOVA; paired

9. Secondary Outcome: Left Ventricular Strain (LVS): Change Immediately Post-Exposure From Baseline
Description: Left ventricular strain will be assessed at baseline prior to exposure (within two weeks), and immediately after the exposure by measuring global longitudinal strain (GLS), an echocardiographic measure of myocardial mechanics. GLS is measured using speckle tracking, a technique by which small myocardial footprints, or speckles, are tracked over the cardiac cycle to enable quantification of left ventricular systolic function. GLS is more sensitive than traditional measures of ventricular function, such as ejection fraction, in detecting clinically inapparent but prognostically important decrements in contractility. The change in global longitudinal strain will be calculated to determine the effect of ozone on left ventricular strain.
Time Frame: Baseline and immediately post-exposure
Population: One participant's LVS data was collected but was not able to undergo analysis due to the shutdown of university laboratories in response to the pandemic
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Filtered Air | Ozone
Number analyzed (Participants) | 13 | 13
percent change | 0.58 (0.44) | 0.06 (0.63)
Statistical Analysis 1: Comparison: Filtered Air vs Ozone; Test type: Superiority; p = 0.50, ANOVA; paired

10. Secondary Outcome: Nasal Epithelial Cell IL-1 Beta Gene Expression: Relative mRNA Counts Immediately Post-Exposure (Baseline-corrected), Ozone vs Filtered Air
Description: RNA isolated from nasal epithelial cell biopsies collected at the screening visit (baseline) within six weeks prior to the first exposure and immediately after each exposure. RNA will be analyzed via real-time quantitative polymerase chain reaction (qPCR) to determine the impact of O3 on inflammatory gene expression.
Time Frame: Screening visit and immediately post-exposure
Population: One participant did not have a pre-exposure nasal epithelial cell biopsy sample available for analysis.
Measure: Mean (Standard Deviation); unit: relative mRNA counts
Arm/Group | Filtered Air | Ozone
Number analyzed (Participants) | 13 | 13
relative mRNA counts | -169.6 (317.5) | -147.4 (329.1)
Statistical Analysis 1: Comparison: Filtered Air vs Ozone; Test type: Superiority; p = 0.54, Wilcoxon signed rank test

11. Secondary Outcome: Flow Mediated Dilation (FMD): Change Immediately Post-Exposure From Baseline
Description: Participants will undergo assesment of flow-mediated brachial artery dilation by brachial ultrasound at baseline prior to exposure (within two weeks), and immediately after exposure to either FA or O3 to assess the impact of O3 exposure on endothelial function. Flow mediated dilation of the brachial artery (FMD) is a noninvasive index of vascular endothelial function. FMD is measured using high-frequency ultrasound, and is expressed as the percent change in arterial diameter in response to the reactive hyperemia induced by 5 minutes of forearm ischemia. Impaired endothelial function leads to atherosclerosis and is associated with an increased risk of cardiovascular events.
Time Frame: Baseline and immediately post-exposure
Population: All participants that completed the study
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Filtered Air | Ozone
Number analyzed (Participants) | 14 | 14
percent change | 1.09 (1.02) | 1.25 (1.04)
Statistical Analysis 1: Comparison: Filtered Air vs Ozone; Test type: Superiority; p = 0.90, ANOVA; paired

12. Secondary Outcome: Change in Heart Rate Variability
Description: Measure was not performed as the equipment (ECG leads and monitor recording heart rate and rhythm) belonged to the EPA and was not made available for this study
Time Frame: baseline, immediately post exposure
Population: No participants analyzed as equipment belonging to the EPA was not available
Arm/Group | Filtered Air | Ozone
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Nasal Epithelial Cell IL-6R Gene Expression: Relative mRNA Counts Immediately Post-Exposure (Baseline-corrected), Ozone vs Filtered Air
Description: as for outcome 10
Time Frame: Screening visit and immediately post-exposure
Population: One participant did not have a pre-exposure nasal epithelial cell biopsy sample available for analysis.
Measure: Mean (Standard Deviation); unit: relative mRNA counts
Arm/Group | Filtered Air | Ozone
Number analyzed (Participants) | 13 | 13
relative mRNA counts | -10.22 (38.5) | -4.72 (25.77)
Statistical Analysis 1: Comparison: Filtered Air vs Ozone; Test type: Superiority; p = 0.64, Wilcoxon signed rank test

14. Secondary Outcome: Nasal Epithelial Cell IL-8 Gene Expression: Relative mRNA Counts Immediately Post-Exposure (Baseline-corrected), Ozone vs Filtered Air
Description: as for outcome 10
Time Frame: Screening visit and immediately post-exposure
Population: One participant did not have a pre-exposure nasal epithelial cell biopsy sample available for analysis.
Measure: Mean (Standard Deviation); unit: relative mRNA counts
Arm/Group | Filtered Air | Ozone
Number analyzed (Participants) | 13 | 13
relative mRNA counts | -537.7 (3470) | 399.7 (5459)
Statistical Analysis 1: Comparison: Filtered Air vs Ozone; Test type: Superiority; p = 0.79, Wilcoxon signed rank test

15. Secondary Outcome: The Percentage of Predicted Forced Vital Capacity (% Predicted FVC): Change Immediately Post-Exposure From Baseline
Description: Participants will be exposed to either filtered air (FA), then ozone (O3), or O3, then FA. Standard spirometry to obtain FEV1 and forced vital capacity (FVC) measurements will be done at baseline within two weeks prior to first exposure, and immediately after exiting the exposure chamber for each exposure. The % Predicted FVC will be calculated from measured versus expected values. The change in % Predicted FVC from baseline to immediately Post-Exposure will be calculated for each participant for each exposure. Values will be compared between FA and O3 to determine the effect of ozone on the % Predicted FVC.
Time Frame: Baseline, immediately post-exposure
Population: All participants that completed the study
Measure: Mean (Standard Deviation); unit: percent predicted FEV1
Arm/Group | Filtered Air | Ozone
Number analyzed (Participants) | 14 | 14
percent predicted FEV1 | -0.3 (0.7) | -1.8 (0.5)
Statistical Analysis 1: Comparison: Filtered Air vs Ozone; Test type: Superiority; p = 0.094, ANOVA

ADVERSE EVENTS:
Time Frame: Up 1 month after completion of the exposures.
Description: Safety assessments included all participants who underwent any study procedures.
Groups:
- Filtered Air: Filtered Air: Participants will be exposed to filtered clean air for 6.5 hours
- Ozone: Ozone: Participants will be exposed to a concentration of ozone for 6.5 hours at a concentration that varies 0.06 to 0.08 PPM
Arm/Group | Filtered Air | Ozone
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 0/15 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-11): https://cdn.clinicaltrials.gov/large-docs/83/NCT02857283/Prot_SAP_000.pdf